CLINICAL TRIAL: NCT04566549
Title: Testing of Hair Products Containing Probiotics
Brief Title: The Safety and Efficacy Evaluation of Hair Products Containing Probiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Chia Nan University of Pharmacy and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: TSMH IRB 20-040-A
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2020-09

CONDITIONS: Skin Problems
Keywords: Hair health; Scalp health; Probiotics; Scalp microbiota
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Shampoo base without probiotics inculding Aqua、Sodium Lauryl Ether Sulphate、Cocamidopropyl Betaine、Cocoamide DEA、Sodium、Polyquaternium-10 、Disodium EDTA、Acrylates Copolymer、Citric Acid、Phenoxyethanol、Fragrance.
  Interventions: Combination Product: Placebo group
- Test group (Active Comparator): Shampoo base with probiotics inculding Aqua、Sodium Lauryl Ether Sulphate、Cocamidopropyl Betaine、Cocoamide DEA、Sodium、Polyquaternium-10 、Disodium EDTA、Acrylates Copolymer、Citric Acid、Phenoxyethanol、Fragrance、Heat-killed Lactobacillus paracasei powders (5x10^8 cells/ g-shampoo).
  Interventions: Combination Product: Test group Probiotic Shampoo

INTERVENTIONS:
Combination Product: Test group Probiotic Shampoo — Probiotic Shampoo
  Other Names: Probiotic Group
  Arms: Test group
Combination Product: Placebo group — Shampoo base
  Other Names: Control Group
  Arms: Placebo group

SUMMARY:
Previous studies on skin health with Lactic acid bacteria (LAB) have been published for many years, including prevention of skin diseases and improvement of skin conditions. In this clinical study, the investigators researched the benefit effects of heat-killed Lactobacillus paracasei shampoo on scalp and hair healthcare.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of hair products containing probiotics

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers between the ages of 20-70.

Exclusion Criteria:

* Subjects are undergoing medical therapy for scalp, hair diseases or diabetes mellitus.
* Subjects with cosmetics allergy.
* Subjects had accepted the scalp surgery such as Follicular Unit Transpalnt, Follicular Unit Extraction in the past half year.
* Subjects with pregnancy or breast-feeding.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Skin Microbiota | Baseline, 4 weeks and 8 weeks
  The changes of scalp microbiota will be evaluated by NGS or qPCR analysis at baseline and different timepoint post-intervention.

SECONDARY OUTCOMES:
The sebum on scalp | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 12 weeks, 20 weeks and 28 weeks
  The scalp sebum will be measured by Sebumeter SM815 (C+K, Germany) at baseline and different timepoint post-intervention.
The scalp flakes (dandruff) | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 12 weeks, 20 weeks and 28 weeks
  The scalp flakes will be evaluated by D-SQAME ® DANDRUFF TESTER at baseline and different timepoint post-intervention.
The hair density (hairs/scalp area) | Baseline, 4 weeks, 8 weeks, 12 weeks, 20 weeks and 28 weeks
  The hair number in a constant scalp area will be measured by Aramo TSII skin/hair diagnosis (Aramhuvis Co., Ltd. Korea) at baseline and different timepoint post-intervention.
Adverse Event | Baseline and 28 weeks
  Any adverse event, such as erythema,rash, itching and so on will be recorded during the intervention.
Single application closed patch epicutaneous test under occlusion | 1 hour, 24 hours and 48 hour
  Probiotics on skin will be evaluated by Human Patch test. The Human Patch test method according to the Guidelines of Human Patch test Standards for Cosmetics, Taiwan Food and Drug Administration, 2019 edition.
Repeated application closed patch epicutaneous test under occlusion | Day 1, 2, 3, 4 and 5
  The irritation potential of probiotics on skin will be evaluated by Human Patch test.
  The Human Patch test method according to the Guidelines of Human Patch test Standards for Cosmetics, Taiwan Food and Drug Administration, 2019 edition.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Gong Lin, PhD, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy and Science, Tainan, Taiwan